CLINICAL TRIAL: NCT07331402
Title: A Random, Single Blind, Positive Control, Crossover Design Clinical Study to Evaluate the Pharmacokinetics and Pharmacodynamics of HSK39004 Inhalation Suspension in COPD Patients
Brief Title: A Clinical Study Evaluating the Pharmacokinetics and Pharmacodynamics of HSK39004 Inhalation Suspension in COPD Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK39004-201
Record Dates: First submitted 2025-08-20; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: COPD Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK39004- Ohtuvayre (Experimental): The first period, HSK39004 inhalation suspension , Inhale through the mouth, 3mg each time, twice a day; The second period，Ohtuvayre inhalation suspension, Inhale through the mouth, 3mg each time, twice a day
  Interventions: Drug: HSK39004 inhalation suspension
- Ohtuvayre - HSK39004 (Other): The first period，Ohtuvayre inhalation suspension, Inhale through the mouth, 3mg each time, twice a day; The second period，HSK39004 inhalation suspension , Inhale through the mouth, 3mg each time, twice a day.
  Interventions: Drug: HSK39004 inhalation suspension

INTERVENTIONS:
Drug: HSK39004 inhalation suspension — HSK39004 inhalation suspension , Inhale through the mouth, 3mg each time, twice a day; Ohtuvayre inhalation suspension, Inhale through the mouth, 3mg each time, twice a day
  Other Names: Ohtuvayre inhalation suspension

SUMMARY:
This is a random, single blind, positive control, crossover design clinical study to evaluate the pharmacokinetics and pharmacodynamics of HSK39004 inhalation suspension in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* During the screening visit (Visit 1), the age range is 40 to 80 years (including the threshold value), and gender is not restricted;
* The subjects with chronic obstructive pulmonary disease (COPD) as per the GOLD 2025 diagnostic criteria, and the symptoms before screening were consistent with COPD for at least 1 year [GOLD 2025 standard: the subjects have chronic respiratory symptoms such as shortness of breath, chronic cough or expectoration, and/or have a history of exposure to risk factors, and the pulmonary function test results show: the forced expiratory volume in one second (FEV1) after using bronchodilators / forced vital capacity (FVC) <0.7];
* During the screening visit (Visit 1):· FEV1/FVC after using bronchodilators is <0.7;· 30% of the expected value ≤ FEV1 after using bronchodilators < 80% of the expected value;
* COPD stable within 4 weeks prior to screening period (Visit 1);
* During the screening period and treatment period, COPD drugs prohibited by the protocol (except for salbutamol inhalation aerosol as a rescue drug) can be discontinued;
* Current smokers with a smoking quantity of ≥ 10 packs per year (smoking index (pack years) = daily smoking quantity (packs) × time (years), 1 pack = 20 cigarettes), or quit smoking for more than 6 months, or those with a history of exposure to other risk factors;
* Participants voluntarily sign the informed consent form；

Exclusion Criteria:

* Have a history of life-threatening COPD, including being admitted to the intensive care unit and/or requiring intubation;
* Have received treatment for COPD acute exacerbation for pneumonia within 12 weeks before screening;
* Have a history of or currently have severe cardiovascular diseases;
* Have type I diabetes or poorly controlled type II diabetes (fasting blood glucose ≥ 10 mmol/L at screening);
* Have cancer (in situ cancer that has been cured for more than 5 years, skin squamous cell carcinoma and basal cell carcinoma, etc., except for subjects with suspected malignant tumors or undetermined tumors);
* Combine other severe unstable kidney, nervous system, endocrine diseases, thyroid diseases, urinary system, ophthalmic diseases, immune system, mental system, gastrointestinal, liver or blood system disease/abnormal history, as determined by the investigator, participation in this study may pose risks to the subjects or affect the analysis of research results;
* During the screening period (visit 1), the investigator determines that the laboratory tests of the subjects show clinically significant abnormalities that may pose risks to the subjects;
* Allergy to HSK39004 inhalation powder or salbutamol or any known components in the administration system ; 8. Before the pulmonary function test during the screening (visit 1), any prohibited drugs in the protocol were used;
* During the screening period, there were clinically significant abnormalities in the 12 lead electrocardiogram that were determined by the researchers to be potentially risky for the subjects;
* Had major surgery (requiring general anesthesia) within 6 weeks before screening, not fully recovered at the time of screening, or planned to undergo surgery before the end of the study;
* Pregnant or lactating women, or female subjects with positive pregnancy test results;
* Researchers determine other subjects who are not suitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The Cmax after single administrations | [Time Frame: From the start of administration to 12 hours post-dose]
  The Cmax of HSK39004 in plasma
The Css(max) after multiple administrations (steady state) | [Time Frame: From the start of administration to 7 days post-dose]
  The Css(max) of HSK39004 in plasma

SECONDARY OUTCOMES:
The ΔFEV1 AUC0-12h | [Time Frame: From the start of administration to 12 hours post-dose on Day1 and Day7]
  The area under the curve of FEV1 change from baseline from 0 to 12 hours after administration
AEs | [Time Frame: From the time of signing ICF to the end of follow-up，up to 7 days after the last administration]
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- 36 Sanhao Street, Heping District, Shenyang, Liaoning,China, Shenyang, Liaoning, China